CLINICAL TRIAL: NCT03896711
Title: MEMORI Corps: A Novel Activity-based Companion Care Program to Benefit Community-living Persons With Dementia, Their Families, and Senior Volunteers
Brief Title: MEMORI Corps: Activity-based Companion Care for Dementia
Acronym: MEMORI Corps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Alzheimer's Association (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00197899; R01AG058586 (NIH)
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Dementia
Keywords: dementia care; community-based; companion care; activity; caregiver wellbeing; caregiver respite; caregiver support; home-based; volunteer
MeSH Terms: conditions — Alzheimer Disease; Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Activity-based companion care program. MEMORI Corps is a companion care model that provides regular companionship and personalized activities to community-living persons with dementia (PWD) delivered by trained volunteer Companion Guides 55 years of age or older. Core intervention components include: (1) detailed virtual assessment of health, well-being, and interests of PWD; (2) personalized activity plans; (3) specialized training of volunteer Companion Guides in virtual program delivery; (4) regular companionship and personalized activities delivered to PWD over 12 weeks; (5) family caregiver education on activity plans and ways to utilize respite opportunities; and (6) multidisciplinary expert support of volunteer companion guides. The goals of the program are to reduce social isolation and improve health and well-being for PWD, reduce burden and support family CGs, and to provide health benefits and meaningful engagement for older volunteer Companion Guides.
Who Masked: Outcomes Assessor
Masking Description: Single blind, pilot, randomized controlled trial where outcome assessors are masked to treatment arm allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Experimental): Intervention arm with MEMORI Corps program
  Interventions: Behavioral: MEMORI Corps program
- Control (Other): Augmented waitlist control.
  Interventions: Other: Augmented Waitlist Control

INTERVENTIONS:
Behavioral: MEMORI Corps program — MEMORI Corps program: Virtual activity-based companion care program. Delivered by trained volunteers 55 years and older, supported by a clinical team, over a 12-week intervention period (up to 5 hours per week, one or more days per week) for each person with dementia/family caregiver dyad. Primary roles of the volunteers are to provide socialization, companionship, and a personalized activity program that focuses on meaningful, engaging and enjoyable activities that match the participant's abilities and interests. Delivered virtually by Zoom.
  Arms: Active Intervention
Other: Augmented Waitlist Control — Participants living with dementia/caregivers will continue any services and supports already engaged with, will receive a free copy of "A Caregiver's Guide to Dementia: Using Activities and Other Strategies to Prevent, Reduce and Manage Behavioral Symptom"), a Resource Guide (ie.,local, regional and national resources), and check-in calls to answer any questions about the materials. Waitlist are offered full intervention after waitlist period. Volunteers randomized to waitlist control continue usual activities (volunteer or other), and resource a resource guide on cognitive health (NIA) and exercise and Physical Activity (Go4Life), referrals to volunteering opportunities, and check-in calls to answer questions and maintain engagement. Waitlist dyads will be followed at specified intervals by the research team and then offered an opportunity for participation in the intervention arm.
  Arms: Control

SUMMARY:
This project adapts a novel activity-based companion care model, the Making Engagement Meaningful through Organized Routine Interaction (MEMORI) Corps intervention, for a virtual delivery format, and then implements the intervention in a pilot, two-arm, randomized controlled trial to evaluate intervention acceptability, feasibility, and preliminary efficacy versus an augmented waitlist control. MEMORI Corps is a companion care model that provides regular companionship and personalized activities to community-living persons with dementia (PWD) delivered by trained volunteer Companion Guides 55 years of age or older. Program goals are to reduce social isolation and improve health and well-being for PWD, reduce burden and provide support to family CGs, as well as provide health benefits and opportunities for meaningful engagement for older volunteer Companion Guides.

DETAILED DESCRIPTION:
This project adapts a novel activity-based companion care model (MEMORI Corps) for community-living persons with dementia for a virtual delivery format, and then implements the intervention in a pilot, two-arm, randomized controlled trial to evaluate intervention acceptability, feasibility, and preliminary efficacy versus an augmented waitlist control. The goals of the program are to reduce social isolation and improve health and well-being for PWD, reduce burden and support family CGs, and to provide health benefits and meaningful engagement for older volunteer Companion Guides.

The target group is 60 dyads (persons living with dementia and their informal co-residing caregiver) and 36 companion guides (health volunteer 55 years of age and older). Participants are randomized 1:1 either to the intervention or waitlist control group. Waitlist participants are offered the opportunity for cross-over into active intervention group. PWD/CG outcomes will be assessed at Baseline, 6-, and 12-weeks (PWD/CG participation lasts 12 weeks). Volunteer Companion Guide outcomes will be assessed at baseline, 6-, and 12-months.

This model program could serve as an important new advancement for community-based long term care for PWD that addresses unmet patient- and family-centered needs through civic engagement of seniors. It could also serve as an intervention for dementia risk-reduction and brain health if found to be efficacious.

Specific aims are to:

Aim 1: Adapt and refine the MEMORI Corps intervention for a virtual delivery format using iterative user-centered design principles and multiple stakeholder input.

Aim 2: Conduct a pilot, two-arm, randomized controlled trial to evaluate acceptability, feasibility, safety, and preliminary efficacy of the MEMORI Corps intervention (vs. wait list control group) in 60 community-living person's living with demential (PLWD) and informal caregiver dyads and 36 volunteer companion guides from geographically and demographically diverse regions in Maryland.

Aim 3: Evaluate the feasibility of ascertainment of community-living PLWD, caregiver, and volunteer-level outcomes over time using virtual and telephonic data collection methods.

ELIGIBILITY:
Inclusion Criteria:

Persons with dementia and informal caregiver (PWD/CG) must both meet eligibility criteria. These criteria are designed to reduce PWD/CG attrition and ensure safety of PWD, CG, and volunteers.

PWD are eligible if:

* English speaking;
* Have an established physician clinical diagnosis of dementia (any stage) and confirmed with Informant Questionnaire on Cognitive Decline in the. Elderly (IQCODE) cut off >=52 ,
* Are able to participate in at least 4 basic Activities of Daily Living (out of 11),
* Have not received formal (i.e., in-home companion care, or adult day center) activity-focused care services in the past 4 weeks,
* Living at home in all counties in Maryland and Baltimore City,
* Have a co-residing informal caregiver willing to participate as study partner, and 30 years old or older.

CG are eligible if:

* English speaking,
* 21 years of age or older (male or female),
* Deemed to be a reliable informal caregiver (not paid for caregiving of PWD) who knows the PWD well,
* Co-residing with the PWD, and
* Relied on by the PWD for assistance in activities of daily living (instrumental or basic).

Volunteers (i.e. "Companion Guides") are eligible if:

* English-speaking,
* 55 years or older, (3) High School diploma or General Equivalency Diploma (GED) (minimum) (2) ability pass a basic adult literacy screen
* Ability to pass a background check, physical and mental health screening,
* A Montreal Cognitive Assessment (MoCA)-Blind score of 18 or above,
* Ability to commit to 12 months of service (5 hours per week, excluding travel time and continuing education and support), and
* Are reliable during intake and on-boarding process and able to successfully complete training.

Exclusion Criteria:

PWD are excluded if:

* Deemed to be in a crisis/unsafe situation at baseline,
* Planned transition from home in less than 6 months,
* At end-stage disease (e.g. bed-bound and non-communicative, or hospice),
* Currently enrolled in a dementia related clinical trial, or
* Deemed to have severe behavioral symptoms so severe that participation in this study is unsafe (e.g., are placing self or others at harm).

CGs are excluded if:

* Do not plan to be co-residing with the PWD in the next 6 months, or
* Currently involved in a behavioral/educational clinical trial.

Volunteers are excluded:

* Planning on moving from the area in the next 12 months,
* Unable to provide informed consent, and
* Report having an existing cognitive disorder diagnosis by a health provider (e.g., Mild Cognitive Impairment, Alzheimer's disease or other type of dementia).

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2025-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quincy Samus, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, we received over 650 community-based referrals from over 20 unique community-based referral sources (including health care and non-health care related sources).
Pre-assignment Details: Completed enrollment of 175 individual participants. 173 were randomized (61 Persons Living With Dementia (PLWD), 61 Family Caregivers, 51 Volunteer/Companion Guides). 1 dyad was inadvertently not randomized after baseline and excluded from analysis.
Groups:
- Active Intervention: Intervention arm with MEMORI Corps program
  MEMORI Corps program: Virtual activity-based companion care program. Delivered by trained senior volunteers, supported by a clinical team, over a 12-week intervention period (up to 5 hours per week, one or more days per week) for each person with dementia/family caregiver dyad. Primary roles of the volunteers are to provide socialization, companionship, and a personalized activity program that focuses on meaningful, engaging and enjoyable activities that match the participant's abilities and interests.
- Control: Augmented waitlist control.
  Augmented Waitlist Control: Persons with dementia/caregivers will continue any services and supports being used, will receive a free copy of "A Caregiver's Guide to Dementia: Using Activities and Other Strategies to Prevent, Reduce and Manage Behavioral Symptom"103), a Resource Guide with written educational materials on local, regional and national resources, management of CG stress/well-being, and check-in calls to answer any questions about the materials. Volunteers randomized to waitlist control will continue with usual activities (volunteer or other), and will receive additional written educational materials on cognitive health (NIA) and exercise and Physical Activity (Go4Life), referrals to the Baltimore City Commission on Aging and Retirement Education for volunteering opportunities, and check-in calls to answer questions and maintain engagement. Waitlist dyads will be followed at specified intervals by the research team and then offered an opportunity for participation in the intervention arm.
Period: Overall Study
Arm/Group | Active Intervention | Control
Started | 90 | 83
PLWD | 33 | 28
Family Caregivers | 33 | 28
Volunteer/Companion Guides | 24 | 27
Completed | 72 | 70
Not Completed | 18 | 13

BASELINE CHARACTERISTICS:
Groups:
- Control: Augmented waitlist control.
  Augmented Waitlist Control: Participants living with dementia/caregivers will continue any services and supports thy are already engaged with, will receive a free copy of "A Caregiver's Guide to Dementia: Using Activities and Other Strategies to Prevent, Reduce and Manage Behavioral Symptom"), a Resource Guide (ie.,local, regional and national resources), and check-in calls to answer any questions about the materials. Waitlist are offered full intervention after waitlist period. Volunteers randomized to waitlist control continue their usual activities (volunteer or other), and resource a resource guide on cognitive health (NIA) and exercise and Physical Activity (Go4Life), referrals to volunteering opportunities, and check-in calls to answer questions and maintain engagement. Waitlist dyads will be followed at specified intervals by the research team and then offered an opportunity for participation in the intervention arm.
- Total: Total of all reporting groups
Arm/Group | Active Intervention | Control | Total
Number analyzed (Participants) | 90 | 83 | 173
Age, Categorical [Count of Participants; unit: Participants] — Population: The total participant sample is comprised of 3 subgroups of participants (Persons living with Dementia, Caregivers, and Volunteer Companion Guides) and these have been represented separately in rows.
  Participants
    Persons living with dementia: number analyzed (Participants) | 33 | 28 | 61
    Persons living with dementia: <=18 years | 0 | 0 | 0
    Persons living with dementia: Between 18 and 65 years | 5 | 3 | 8
    Persons living with dementia: >=65 years | 28 | 25 | 53
    Dementia Caregivers: number analyzed (Participants) | 33 | 28 | 61
    Dementia Caregivers: <=18 years | 0 | 0 | 0
    Dementia Caregivers: Between 18 and 65 years | 11 | 12 | 23
    Dementia Caregivers: >=65 years | 22 | 16 | 38
    Volunteer Companion Guides: number analyzed (Participants) | 24 | 27 | 51
    Volunteer Companion Guides: <=18 years | 0 | 0 | 0
    Volunteer Companion Guides: Between 18 and 65 years | 10 | 12 | 22
    Volunteer Companion Guides: >=65 years | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The total participant sample is comprised of 3 subgroups of participants (Persons living with Dementia, Caregivers, and Volunteer Companion Guides) and these have been represented separately in rows.
  years
    Persons living with dementia: number analyzed (Participants) | 33 | 28 | 61
    Persons living with dementia | 78.03 (8.95) | 75.46 (8.50) | 76.85 (8.77)
    Dementia Caregivers: number analyzed (Participants) | 33 | 28 | 61
    Dementia Caregivers | 69.18 (9.12) | 64.64 (9.99) | 67.10 (9.72)
    Volunteer Companion Guides: number analyzed (Participants) | 24 | 27 | 51
    Volunteer Companion Guides | 66.58 (7.78) | 65.78 (8.17) | 66.16 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The total participant sample is comprised of 3 subgroups of participants (Persons living with Dementia, Caregivers, and Volunteer Companion Guides) and these have been represented separately in rows.
  Participants
    Person Living with Dementia: number analyzed (Participants) | 33 | 28 | 61
    Person Living with Dementia: Female | 13 | 13 | 26
    Person Living with Dementia: Male | 20 | 15 | 35
    Dementia Caregiver: number analyzed (Participants) | 33 | 28 | 61
    Dementia Caregiver: Female | 25 | 23 | 48
    Dementia Caregiver: Male | 8 | 5 | 13
    Volunteer Companion Guide: number analyzed (Participants) | 24 | 27 | 51
    Volunteer Companion Guide: Female | 22 | 23 | 45
    Volunteer Companion Guide: Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The total participant sample is comprised of 3 subgroups of participants (Persons living with Dementia, Caregivers, and Volunteer Companion Guides) and these have been represented separately in rows.
  Participants
    Person Living with Dementia: number analyzed (Participants) | 33 | 28 | 61
    Person Living with Dementia: American Indian or Alaska Native | 0 | 0 | 0
    Person Living with Dementia: Asian | 0 | 0 | 0
    Person Living with Dementia: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Person Living with Dementia: Black or African American | 11 | 11 | 22
    Person Living with Dementia: White | 22 | 17 | 39
    Person Living with Dementia: More than one race | 0 | 0 | 0
    Person Living with Dementia: Unknown or Not Reported | 0 | 0 | 0
    Dementia Caregiver: number analyzed (Participants) | 33 | 28 | 61
    Dementia Caregiver: American Indian or Alaska Native | 0 | 0 | 0
    Dementia Caregiver: Asian | 0 | 1 | 1
    Dementia Caregiver: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Dementia Caregiver: Black or African American | 11 | 12 | 23
    Dementia Caregiver: White | 22 | 14 | 36
    Dementia Caregiver: More than one race | 0 | 1 | 1
    Dementia Caregiver: Unknown or Not Reported | 0 | 0 | 0
    Volunteer Companion Guide: number analyzed (Participants) | 24 | 27 | 51
    Volunteer Companion Guide: American Indian or Alaska Native | 0 | 1 | 1
    Volunteer Companion Guide: Asian | 0 | 0 | 0
    Volunteer Companion Guide: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Volunteer Companion Guide: Black or African American | 8 | 3 | 11
    Volunteer Companion Guide: White | 14 | 22 | 36
    Volunteer Companion Guide: More than one race | 2 | 1 | 3
    Volunteer Companion Guide: Unknown or Not Reported | 0 | 0 | 0
Neuropsychiatric Inventory (NPI) Score [Mean (Standard Deviation); unit: units on a scale] — Person with dementia measure. The total score (frequency x severity) of the Neuropsychiatric Inventory (NPI) scale will be used to measure neuropsychiatric and behavioral symptoms. The NPI is a proxy rating of person with dementia's severity, frequency, and distress across 12 types of neuropsychiatric behavior problems. Scores can range from 0-144, with higher score indicating greater neuropsychiatric behavioral burden. Population: This baseline measure is for a subset of participants (i.e., persons living with dementia, PWD). Excludes caregiver and senior volunteer companion guide participants.
  units on a scale
    number analyzed (Participants) | 33 | 28 | 61
    (all) | 21.80 (19.36) | 17.38 (14.79) | 19.51 (19.50)
Quality of Life in Alzheimer's Disease (QOL-AD) [Mean (Standard Deviation); unit: units on a scale] — The total score (sum of all items) for the Quality of life in Alzheimer's Disease (QOL-AD) tool will assess quality of life in the context of Alzheimer's Disease. The QOL-AD has a self-rated and proxy-rated version for persons with dementia, and was specifically developed for use in dementia. Scores can range from 13-52, with higher scores indicating better quality of life. Population: This baseline measure is for a subset of participants (i.e., persons living with dementia, PWD). Excludes caregiver and senior volunteer companion guide participants.
  units on a scale
    number analyzed (Participants) | 33 | 28 | 61
    (all) | 33.54 (6.29) | 31.22 (4.01) | 32.67 (5.78)
Zarit Burden Inventory-Short Form [Mean (Standard Deviation); unit: units on a scale] — The total score (sum of items) for the Zarit Burden Inventory-Short Form-12 items (ZBI) will assess subjective caregiver burden. The ZBI short form is a self-rated 12-item measure of caregiver subjective burden rating related to caregiving for persons with dementia. Scores can range from 0-48, with higher scores indicating greater perceived burden. Population: This baseline measure is for a subset of participants (i.e., Caregivers of persons living with dementia-CGs). Excludes persons living with dementia and senior volunteer companion guide participants.
  units on a scale
    number analyzed (Participants) | 33 | 28 | 61
    (all) | 16.51 (7.70) | 19.56 (6.57) | 17.72 (7.36)
Patient Health Questionnaire (PHQ) - 8 [Mean (Standard Deviation); unit: units on a scale] — The total score (sum of items) for the The Patient Health Questionnaire (PHQ) - 8 will assess depressive symptoms severity. The PHQ-8 is a self-rated 8 item measure of caregiver depressive symptoms. Scores can range from 0-24, with higher scores indicating greater depressive symptoms. Population: This baseline measure is for a subset of participants (i.e., persons living with dementia, PWD). Excludes caregiver and senior volunteer companion guide participants.
  units on a scale
    number analyzed (Participants) | 33 | 28 | 61
    (all) | 4.08 (4.49) | 4.18 (5.03) | 4.14 (4.69)
Leisure Activity Participation Impact Scale [Mean (Standard Deviation); unit: units on a scale] — 11 item scale measuring the subjective impact of leisure activity participation on several areas of life and emotional well-being. Scores range from 11-55 with higher scores indicating more beneficial subjective impact of leisure activities Population: This baseline measure is for a subset of participants (i.e., persons living with dementia, PWD). Excludes caregiver and senior volunteer companion guide participants.
  units on a scale
    number analyzed (Participants) | 33 | 28 | 61
    (all) | 42.21 (7.51) | 40.45 (5.47) | 41.66 (6.80)
UCLA 3 Loneliness Scale [Mean (Standard Deviation); unit: units on a scale] — Three item measure of perceived loneliness and social isolation. Scores range from 3-9 with higher scores indicating higher levels of loneliness. Population: This baseline measure is for a subset of participants (i.e., persons living with dementia, PWD). Excludes caregiver and senior volunteer companion guide participants.
  units on a scale
    number analyzed (Participants) | 33 | 28 | 61
    (all) | 4.65 (1.80) | 4.05 (1.60) | 4.36 (1.69)
Caregiver UCLA 3 Loneliness Scale [Mean (Standard Deviation); unit: units on a scale] — Three item measure of perceived loneliness and social isolation. Scores range from 3-9 with higher scores indicating higher levels of loneliness. Population: This baseline measure is for a subset of participants (i.e., caregivers of persons living with dementia). Excludes persons living with dementia and senior volunteer companion guide participants.
  units on a scale
    number analyzed (Participants) | 33 | 28 | 61
    (all) | 4.71 (1.82) | 5.00 (1.72) | 4.81 (1.77)
Caregiver Time Spent Helping PLWD in Last Week [Mean (Standard Deviation); unit: hours per week] — This item ask caregivers to estimate hours spent in past week helping or doing activities for the person living with dementia. Higher values indicate greater number of hours spent helping or doing activities for with the person living with dementia. Population: This baseline measure is for a subset of participants (i.e., caregivers of PWD). Excludes person with dementia (PWD) and senior volunteer companion guide participants.
  hours per week
    number analyzed (Participants) | 33 | 28 | 61
    (all) | 50.84 (47.07) | 49.48 (43.38) | 50.22 (45.04)
Senior Companion Volunteers Patient Health Questionnaire ( [Mean (Standard Deviation); unit: units on a scale] — The total score (sum of items) for the The Patient Health Questionnaire (PHQ) - 8 will assess depressive symptoms severity in senior companion volunteers. The PHQ-8 is a self-rated 8 item measure of caregiver depressive symptoms. Scores can range from 0-24, with higher scores indicating greater depressive symptoms. Population: This baseline measure is for a subset of participants (i.e., senior volunteer companion guide participants). Excludes persons living with dementia and caregiver participants.
  units on a scale
    number analyzed (Participants) | 24 | 27 | 51
    (all) | 1.54 (1.61) | 1.46 (1.88) | 1.49 (1.71)

OUTCOME MEASURES:

1. Primary Outcome: Change in Neuropsychiatric Symptoms as Assessed by Neuropsychiatric Inventory (NPI) Score
Description: The total score (frequency x severity) of the Neuropsychiatric Inventory (NPI) scale will be used to measure neuropsychiatric and behavioral symptoms. The NPI is a proxy rating of person with dementia's severity, frequency, and distress across 12 types of neuropsychiatric behavior problems. Scores can range from 0-144, with higher score indicating greater neuropsychiatric behavioral burden.
Time Frame: Baseline - 12 weeks
Population: Person with dementia participant outcome, intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 26 | 19
score on a scale | 3.35 (11.14) | 0.47 (6.10)

2. Primary Outcome: Change in Quality of Life as Assessed by the Quality of Life in Alzheimer's Disease (QOL-AD) Tool
Description: The total score (sum of all items) for the Quality of life in Alzheimer's Disease (QOL-AD) tool will assess quality of life in the context of Alzheimer's Disease. The QOL-AD has a self-rated and proxy-rated version for persons with dementia, and was specifically developed for use in dementia. Scores can range from 13-52, with higher scores indicating better quality of life.
Time Frame: Baseline - 12 weeks
Population: Person with dementia participant outcome, intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 19 | 18
units on a scale | 0.21 (3.44) | -0.44 (4.97)

3. Primary Outcome: Change in Subjective Caregiver Burden as Assessed by the Zarit Burden Inventory-Short Form
Description: The total score (sum of items) for the Zarit Burden Inventory-Short Form-12 items (ZBI) will assess subjective caregiver burden. The ZBI short form is a self-rated 12-item measure of caregiver subjective burden rating related to caregiving for persons with dementia. Scores can range from 0-48, with higher scores indicating greater perceived burden.
Time Frame: Baseline - 12 weeks
Population: Caregivers of persons with dementia participants, Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 26 | 23
units on a scale | 0.04 (4.84) | -0.69 (5.84)

4. Primary Outcome: Change in Depressive Symptoms in Caregivers as Assessed by The Patient Health Questionnaire (PHQ) - 8
Description: The total score (sum of items) for the The Patient Health Questionnaire (PHQ) - 8 will assess depressive symptoms severity. The PHQ-8 is a self-rated 8 item measure of caregiver depressive symptoms. Scores can range from 0-24, with higher scores indicating greater depressive symptoms.
Time Frame: Baseline - 12 weeks
Population: Caregiver of person living with dementia outcome, intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 26 | 22
units on a scale | 0.38 (3.97) | 0.59 (2.97)

5. Primary Outcome: Change in Perceived Loneliness as Measured by UCLA 3 Loneliness Scale
Description: Three item measure of perceived loneliness and social isolation. Scores range from 3-9 with higher scores indicating higher levels of loneliness.
Time Frame: Baseline - 12 weeks
Population: Person living with dementia participant outcome, intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 15 | 19
units on a scale | 0.20 (1.86) | -0.42 (1.07)

6. Primary Outcome: Change in Perceived Loneliness for Caregiver as Measured by UCLA 3 Loneliness Scale
Description: as for outcome 5
Time Frame: Baseline - 12 weeks
Population: Caregiver of person with dementia outcome, intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 23 | 20
units on a scale | -0.39 (1.23) | 0.10 (1.71)

7. Primary Outcome: Program Satisfaction and Perceived Impact Survey
Description: 55 item likert scale survey assessing program delivery, feasibility, acceptability, perceived program impact. Total score range from 55-253 with higher scores indicating greater satisfaction and perceived feasibility, with higher scores indicating
Time Frame: 12-weeks post intervention
Population: caregivers in intervention arm only of persons with dementia receiving intervention, intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 26 | 0
score on a scale | 124.15 (25.20) |

8. Primary Outcome: Change in Perceived Impact of Leisure Activities as Measured by Leisure Activity Participation Impact Scale
Description: 11 item scale measuring the subjective impact of leisure activity participation on several areas of life and emotional well-being. Scores range from 11-55 with higher scores indicating more beneficial subjective impact of leisure activities
Time Frame: Baseline - 12 weeks
Population: Person living with dementia participant outcome, intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 21 | 16
score on a scale | -1.71 (4.01) | -1.63 (4.46)

9. Secondary Outcome: Change in Caregiver Time Spent Helping Person Living With Dementia
Description: Two individual items ask caregivers to estimate hours per day spent doing caregiving activities, and hours per day spent with the person with dementia in a typical week. Objective measure of caregiver burden. Higher time estimates in performing these tasks indicate greater objective burden.
Time Frame: Baseline - 12 weeks
Population: caregiver of person living with dementia participant outcomes, intent to treatment
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 26 | 23
hours per week | -14.04 (45.56) | -0.96 (29.37)

10. Secondary Outcome: Change in Depressive Symptoms in Senior Companion Volunteers as Assessed by The Patient Health Questionnaire (PHQ) - 8
Description: The total score (sum of items) for the The Patient Health Questionnaire (PHQ) - 8 will assess depressive symptoms severity in senior companion volunteers. The PHQ-8 is a self-rated 8 item measure of caregiver depressive symptoms. Scores can range from 0-24, with higher scores indicating greater depressive symptoms.
Time Frame: Baseline -12 weeks
Population: Outcome is only for senior companion guide volunteer participants, intent to treat. This outcome is for a subset of participants (i.e., senior volunteer companion guides). Excludes PLWD and caregiver participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Intervention | Control
Number analyzed (Participants) | 24 | 27
units on a scale | 1.02 (2.61) | 0.80 (1.79)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks for persons living with dementia. Up to 24 months for healthy volunteer companion guide participants.
Description: Adverse event data was not collected for family caregivers.
Groups:
- Active Intervention-PLWD; Active Intervention - Volunteer/Companion Guides: Intervention arm with MEMORI Corps program
  MEMORI Corps program: Virtual activity-based companion care program. Delivered by trained senior volunteers, supported by a clinical team, over a 12-week intervention period (up to 5 hours per week, one or more days per week) for each person with dementia/family caregiver dyad. Primary roles of the volunteers are to provide socialization, companionship, and a personalized activity program that focuses on meaningful, engaging and enjoyable activities that match the participant's abilities and interests.
- Waitlist Control - PLWD; Waitlist Control - Volunteer/Companion Guides; Waitlist Received Intervention - Volunteer/Companion Guides: tervention arm with MEMORI Corps program
  MEMORI Corps program: Virtual activity-based companion care program. Delivered by trained senior volunteers, supported by a clinical team, over a 12-week intervention period (up to 5 hours per week, one or more days per week) for each person with dementia/family caregiver dyad. Primary roles of the volunteers are to provide socialization, companionship, and a personalized activity program that focuses on meaningful, engaging and enjoyable activities that match the participant's abilities and interests.
- Waitlist Received Intervention - PLWD: Augmented waitlist control.
  Augmented Waitlist Control: Persons with dementia/caregivers will continue any services and supports being used, will receive a free copy of "A Caregiver's Guide to Dementia: Using Activities and Other Strategies to Prevent, Reduce and Manage Behavioral Symptom"103), a Resource Guide with written educational materials on local, regional and national resources, management of CG stress/well-being, and check-in calls to answer any questions about the materials. Volunteers randomized to waitlist control will continue with usual activities (volunteer or other), and will receive additional written educational materials on cognitive health (NIA) and exercise and Physical Activity (Go4Life), referrals to the Baltimore City Commission on Aging and Retirement Education for volunteering opportunities, and check-in calls to answer questions and maintain engagement. Waitlist dyads will be followed at specified intervals by the research team and then offered an opportunity for participation in the intervention arm.
Arm/Group | Active Intervention-PLWD | Active Intervention - Volunteer/Companion Guides | Waitlist Control - PLWD | Waitlist Control - Volunteer/Companion Guides | Waitlist Received Intervention - PLWD | Waitlist Received Intervention - Volunteer/Companion Guides
All-Cause Mortality (participants affected / at risk) | 0/33 | 1/24 | 0/28 | 0/27 | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/24 | 0/28 | 0/27 | 0/22 | 0/5
Other Adverse Events (participants affected / at risk) | 0/33 | 0/24 | 0/28 | 0/27 | 0/22 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT03896711/Prot_SAP_000.pdf